CLINICAL TRIAL: NCT05985525
Title: Microvascular Monitoring in Circulatory Shock and Sepsis (MiMICSS): Prospective Observational Cohort Study
Brief Title: Microvascular Monitoring in Circulatory Shock and Sepsis (MiMICSS)
Acronym: MiMICSS
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Asher Mendelson, Assistant Professor, University of Manitoba
Other Study IDs: HS25043
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Shock; Critical Illness
Keywords: Near-Infrared Spectroscopy
MeSH Terms: conditions — Sepsis; Shock; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: All patients
  Interventions: Device: Skeletal muscle and cerebral NIRS (research device)

INTERVENTIONS:
Device: Skeletal muscle and cerebral NIRS (research device) — NIRS applied on skeletal muscle and brain on days 1, 3, and 8 of ICU admission. Monitoring applied for up to 24hrs on each day.
  Other Names: PortaMon (Artinis Inc, Netherlands); PortaLite (Artinis Inc, Netherlands)

SUMMARY:
Investigation of the feasibility of using near-infrared spectroscopy (NIRS) to monitor microvascular function in critically ill patients.

DETAILED DESCRIPTION:
This is a prospective observational study using non-invasive NIRS for microvascular monitoring in the ICU. The study involves no interventions above standard of care other than the application of the NIRS monitors.

NIRS will be applied to skeletal muscle and the brain longitudinally throughout ICU admission. Vital signs are extracted continuously from the ICU monitor and clinical data are recorded from patient records.

The broad goals of the study are:

1. Determine the feasibility of longitudinal NIRS monitoring in ICU patients
2. Determine the ability to derive patient-specific microvascular metrics using NIRS
3. Explore the relationship between microvascular metrics and ICU mortality

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ICU
* Receiving invasive mechanical ventilation

Exclusion Criteria:

* Body Mass Index >40
* More than 24 hours has elapsed since ICU admission
* Death is deemed to be imminent and inevitable during the next 24 hours
* Known allergy to the textile components of the device
* Significant clinical jaundice, ecchymosis
* COVID positive microbiological result
* The treating clinician believes that participation in the domain would not be in the best interests of the patient
* Consent declined from patient or authorized third party

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted to the ICU receiving invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 30 days
  Recruitment of two patients per month from each study site

SECONDARY OUTCOMES:
protocol adherence | 14 days
  collection of NIRS and clinical data for each monitoring session
NIRS and vital sign data quality | 14 days
  NIRS and vital sign data is >50% free of artifacts for >80% of recording sessions to enable further analysis
Optimal Map (MAPopt) derivation | 14 days
  when MAP and NIRS data available together, ability to derive MAPopt from >80% of recording sessions using correlation analysis

OTHER OUTCOMES:
ICU mortality | 30 days
  ICU mortality status
Hospital mortality | 100 days
  Hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Asher Mendelson, MD, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre Winnipeg, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No